CLINICAL TRIAL: NCT02193347
Title: Patients With IDH1 Positive Recurrent Grade II Glioma Enrolled in a Safety and Immunogenicity Study of Tumor-Specific Peptide Vaccine
Brief Title: IDH1 Peptide Vaccine for Recurrent Grade II Glioma
Acronym: RESIST
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Katy Peters, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Katy Peters, MD, PhD, Associate Professor, Neurology and Neurosurgery, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00054746
Record Dates: First submitted 2014-07-02; First posted 2014-07-17 (Estimated); Results first posted 2021-03-15 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-02

CONDITIONS: Brain Cancer; Brain Neoplasm, Primary; Brain Neoplasms, Recurrent; Brain Tumor; Cancer of the Brain
Keywords: Immunotherapy; Adult
MeSH Terms: conditions — Brain Neoplasms; Recurrence | interventions — Diphtheria-Tetanus Vaccine; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PEPIDH1M vaccine (Experimental): PEPIDH1M vaccine is made up of a peptide that spans the mutated region of IDH1R132H (Isocitrate Dehydrogenase 1). The peptide is administered with GM-CSF (Granulocyte Macrophage Colony Stimulating Factor) mixed with Montanide ISA 51.
  Interventions: Biological: PEPIDH1M vaccine; Biological: Tetanus-Diphtheria Toxoid (Td); Drug: Temozolomide

INTERVENTIONS:
Biological: PEPIDH1M vaccine — PEPIDH1M vaccine is made up of 500 µg of 25 amino acid peptide administered with 150 µg of GM-CSF mixed 1:1 with Montanide ISA 51 administered intradermally. The peptide vaccine is administered in the groin area approximately 10 cm below the inguinal ligament.
Biological: Tetanus-Diphtheria Toxoid (Td) — After consent has been signed, all subjects will undergo standard of care vaccination with 0.5 mL of Td (tetanus and diphtheria toxoids adsorbed) intramuscularly (I.M.) into the deltoid muscle to ensure adequate immunity to the tetanus antigen. Within 48 hours of leukapheresis, subjects will receive a vaccine site pre-conditioning as a single dose of Td toxoid (1 flocculation unit, Lf, in a total volume of 0.4 mLs saline) administered intradermally to the right side of the groin one day prior to receiving the first PEPIDH1M vaccine.
  Other Names: Tenivac
Drug: Temozolomide — Subjects are treated with temozolomide (TMZ) at a targeted dose of 50-100mg/m2/d for 21 days every 28 days for up to 12 cycles. Subjects that have transitioned to a higher grade brain tumor at time of surgery will receive TMZ and radiation therapy per standard of care before starting TMZ cycles.
  Other Names: Temodar

SUMMARY:
Potential subjects with progressive Grade II primary brain tumor that have IDH1 positive testing from the primary tumor (initial diagnosis) will be offered this treatment study in order to test the safety of the PEPIDH1M vaccine in combination with standard chemotherapy (temozolomide).

DETAILED DESCRIPTION:
After informed consent has been signed, subjects will undergo standard of care vaccination with 0.5 mL of Td (tetanus and diphtheria toxoids adsorbed) intramuscularly into the deltoid muscle to ensure adequate immunity to the tetanus antigen.

Eligible subjects will undergo a 1-2 hour leukapheresis (to pull off white blood cells) for immune monitoring. Within 48 hours of leukapheresis, subjects will receive vaccine site pre-conditioning as a single dose of Td toxoid (in a total volume of 0.4 mLs salt water/saline) given in the intradermal space (just under the surface of the skin) to the right groin area. The pre-conditioning will be administered one day prior to receiving PEPIDH1M vaccine. The peptide vaccine is administered in the upper thigh area approximately 4 inches below the groin in the intradermal space as vaccine # 1. Subsequent vaccines will be given on day 15 ±3 days (vaccine #2) and day 29 ±3 days (vaccine #3). Each injection of the peptide vaccine will be given half on the right groin and half on the left groin. The first 3 peptide vaccine injections will occur without temozolomide (standard of care chemotherapy).

Seven to twelve days after the 3rd vaccine, subjects will have standard of care surgery to remove the tumor. Tumor samples will be evaluated for the IDH1 markers and analyzed for other cells that may have entered the tumor.

Based on the the tissue obtained at surgery, subjects with stable histologic grade at recurrence will then be treated with vaccine and temozolomide. During monthly cycles of temozolomide, subjects will receive the vaccine on day 22 (+ 2 days) for a maximum of 15 total vaccines (which includes the first 3 bi-weekly vaccines). Patients that have transitioned to a higher grade brain tumor at the time of surgery will receive temozolomide and radiation therapy per standard of care and monthly vaccines (vaccines #4-6). After completion of radiation therapy, subjects in this treatment group will receive vaccines monthly on day 22 (+2 days) with post-RT cycles of TMZ to a maximum of 15 vaccines.

All Adverse Events will be collected from time of consent until off study. The treatment phase of the study will end 1 month after the last vaccine. Patients will be followed only for overall survival, progression-free survival, and subsequent therapies thereafter.

Subjects will have blood collected for immune monitoring and biomarker testing during the following times: prior to initiating vaccine therapy (at the leukapheresis visit), prior to surgery to remove the tumor, at the clinic visit prior to starting first cycle of temozolomide after surgery (or radiation therapy and temozolomide for those who transition to higher grade), at vaccine #6, and at end of vaccine treatment (1 month after vaccine #15 or time the subject comes off study, whichever comes first).

Subjects will be imaged with contrast-enhanced magnetic resonance imaging (MRI) according to standard of care every 10 weeks (+/- 4 weeks) while on temozolomide and afterward, per the treating neuro-oncologist's recommendation. Revised Assessment in Neuro-Oncology (RANO) criteria will be used for assessment of pseudoprogression and tumor progression. Subjects demonstrating definitive progression will be removed from study.

As part of standard care for these subjects, upon tumor progression, participants may undergo biopsy or resection. As this is not a research procedure, consent will be obtained separately. Subjects that have this procedure done within the Duke University Health System will be asked to have a portion of the tumor sample, if possible, to assess immunologic cell infiltration, antigen expression, and biomarkers for immunologic response.

Please note, data collection will continue to occur outside of the defined primary and secondary outcomes for exploratory objectives.

The specific exploratory objective involves describing the progression free survival (PFS) and overall survival (OS). The endpoint is the proportion of patients alive without disease progression 6 months after initial vaccine treatment, and both the median PFS, and the median OS.

The objective will be reviewed at 3 years after the last subject came off study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. IDH1R132H expression in primary tumor
3. Radiographic and/or clinical progressive and resectable Grade II glioma.
4. Signed informed consent.
5. For females of child-bearing potential, negative serum pregnancy test at screening (within 48 hours prior to leukapheresis)
6. Women of childbearing potential and male participants must agree to practice adequate contraception.
7. Karnofsky Performance Status (KPS) of ≥ 70.
8. Complete Blood Count (CBC)/differential with adequate bone marrow function as defined below within 2 weeks of enrollment:

   * Absolute neutrophil count, ≥ 1500 cells/mm3.
   * Platelet count, ≥ 100,000 cells/mm3.
   * Hemoglobin ≥ 10 g/dl. (Note: the use of transfusion or other intervention to achieve Hgb ≥ 10 g/dl is acceptable.)
9. Adequate renal function as defined below within 2 weeks of enrollment:

   * Blood Urea Nitrogen (BUN) ≤ 25 mg/dl.
   * Creatinine ≤ 1.7 mg/dl.
10. Adequate hepatic function as defined below within 2 weeks of enrollment:

    * Bilirubin ≤ 2.0 mg/dl.
    * Alanine Aminotransferase (ALT) ≤ 3 x normal range.
    * Aspartate Aminotransferase (AST) ≤ 3 x normal range

Exclusion Criteria:

1. Prior invasive malignancy (except for non-melanomatous skin cancer) unless disease free for ≥ 3 years. (For example, carcinoma in situ of the breast, oral cavity, and cervix are all permissible.)
2. Metastases detected below the tentorium or beyond the cranial vault.
3. Severe, active co-morbidity, defined as follows:

   * Unstable angina and/or congestive heart failure requiring hospitalization.
   * Myocardial infarction within the last 6 months.
   * Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because treatments involved in this protocol may be significantly immunosuppressive.
   * Major medical illnesses or psychiatric impairments that in the investigator's opinion will prevent administration or completion of protocol therapy.
4. Pregnant or lactating women, due to possible adverse effects on the developing fetus or infant due to study drug.
5. Prior allergic reaction to temozolomide.
6. Patients treated on any other therapeutic clinical protocols within 30 days prior to study entry or during participation in the study.
7. Patients with known hypersensitivity to GM-CSF, yeast-derived products, or any component of Leukine®.
8. Allergy or hypersensitivity to tetanus vaccine or any component of the tetanus vaccine.
9. Unable to undergo MRI imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-01-28 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2020-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Peters, M.D., Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PEPIDH1M Vaccine
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PEPIDH1M Vaccine
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.83 (11.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Unacceptable Toxicity
Description: The percentage of patients who experience an unacceptable toxicity defined as any Grade 3 toxicity at least possibly attributed to the vaccine (or vaccine + TMZ and/or RT) that does not resolve to baseline within 3 weeks, any Grade 3 hypersensitivity reactions requiring steroids, any Grade 4 toxicity, including neurologic events not due to progressive disease, or any life threatening-event not attributable to concomitant medication, co-morbid event, or disease progression.
Time Frame: Date of consent through 2 months after the last vaccination
Measure: Number; unit: percentage of participants
Arm/Group | PEPIDH1M Vaccine
Number analyzed (Participants) | 24
percentage of participants | 0

2. Secondary Outcome: Percentage of Patients With a Positive Vaccine Response After 3 Post-Surgery Vaccines as Measured by IFNγ ELIspot
Description: Assess the immunogenicity of the PEPIDH1M vaccine with adjuvant TMZ using ELISpot. This will be done by finding the difference between the number of SFC after 3 post-surgery vaccines and the number of SFC at baseline for each evaluable subject. Immunogenicity will then be summarized by the percentage of evaluable subjects who have a positive vaccine response after 3 post-surgery vaccines. A response will be considered positive if the difference in SFC measurement is greater than 20 SFC per 10^6 lymphocytes after determining the level of detection in the IDH ELISpot.
Time Frame: From time of pheresis #1, one day prior to first pre-surgery vaccine dose, until the time of the third post-surgery vaccination, an expected average of 24 weeks after study initiation
Population: Only 21 of the 24 overall study patients made it far enough on the study to receive 3 post-surgery vaccines and become evaluable for this outcome.
Measure: Number; unit: Percentage of evaluable participants
Arm/Group | PEPIDH1M Vaccine
Number analyzed (Participants) | 21
Percentage of evaluable participants | 42.86

ADVERSE EVENTS:
Time Frame: Date of consent through 2 months after the last vaccination
Arm/Group | PEPIDH1M Vaccine
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 4/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PEPIDH1M Vaccine (N=24)
Anemia (Blood and lymphatic system disorders) | 1
Ventricular arrhythmia (Cardiac disorders) | 1
Other, Specify: CELLULITIS (Infections and infestations) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 2
White blood cell decreased (Investigations) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PEPIDH1M Vaccine (N=24)
Anemia (Blood and lymphatic system disorders) | 20
Sinus tachycardia (Cardiac disorders) | 1
Other, Specify: "INNER EAR PRESSURE" (Ear and labyrinth disorders) | 1
Other, Specify: BLOOD TINGED DRAINAGE (Ear and labyrinth disorders) | 1
Other, Specify: CLICKING SOUND IN LEFT EAR (Ear and labyrinth disorders) | 1
Other, Specify: HEARS CLINKING SOUND IN HEAD INTERMITTENTLY (Ear and labyrinth disorders) | 1
Blurred vision (Eye disorders) | 3
Dry eye (Eye disorders) | 2
Other, Specify: INTERMITTENT PAIN, TWITCHING, AND/OR NUMBNESS UNDER RIGHT EYE (Eye disorders) | 1
Other, Specify: INTERMITTENT; OBJECTS APPEAR TO MOVE OR SHAKE WHEN HOLDING (Eye disorders) | 1
Other, Specify: L EYELID EDEMA (Eye disorders) | 1
Other, Specify: SEEING A "BROWNISH TINTED VERTICAL STRIPE" FROM RIGHT EYE (Eye disorders) | 1
Other, Specify: TUNNEL VISION (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Floaters (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 11
Diarrhea (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 4
Chills (General disorders) | 1
Edema face (General disorders) | 1
Fatigue (General disorders) | 13
Fever (General disorders) | 1
Flu like symptoms (General disorders) | 3
Gait disturbance (General disorders) | 1
Infusion related reaction (General disorders) | 1
Injection site reaction (General disorders) | 24
Pain (General disorders) | 5
Allergic reaction (Immune system disorders) | 1
Bronchial infection (Infections and infestations) | 1
Other, Specify: CELLULITIS (Infections and infestations) | 1
Other, Specify: COLD SORES (Infections and infestations) | 1
Other, Specify: HEAD INCISION WITH DRAINAGE AND TENDERNESS; 2+ SERRATIA MARCESCENS (Infections and infestations) | 1
Other, Specify: INCISION, ABNORMAL TISSUE CULTURE (Infections and infestations) | 1
Other, Specify: SHINGLES (Infections and infestations) | 1
Other, Specify: WOUND INFECTION (Infections and infestations) | 1
Mucosal infection (Infections and infestations) | 1
Papulopustular rash (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Upper respiratory infection (Infections and infestations) | 6
Urinary tract infection (Infections and infestations) | 2
Wound infection (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Other, Specify: LEFT WRIST WOUND (Injury, poisoning and procedural complications) | 1
Other, Specify: LOWER BACK INJURY (Injury, poisoning and procedural complications) | 1
Other, Specify: MVA (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 9
Alkaline phosphatase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 9
Blood bilirubin increased (Investigations) | 3
Creatinine increased (Investigations) | 4
Lymphocyte count decreased (Investigations) | 5
Neutrophil count decreased (Investigations) | 5
Platelet count decreased (Investigations) | 6
White blood cell decreased (Investigations) | 7
Anorexia (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 19
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 6
Hypocalcemia (Metabolism and nutrition disorders) | 12
Hypoglycemia (Metabolism and nutrition disorders) | 6
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 7
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 3
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Other, Specify: BUMPS ON R FOREARM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Other, Specify: L WRIST BUMP/NODULE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Concentration impairment (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 7
Dysgeusia (Nervous system disorders) | 1
Dysphasia (Nervous system disorders) | 8
Facial nerve disorder (Nervous system disorders) | 1
Headache (Nervous system disorders) | 10
Memory impairment (Nervous system disorders) | 5
Movements involuntary (Nervous system disorders) | 1
Other, Specify: AURA (Nervous system disorders) | 1
Other, Specify: DECREASED CIRCULATION IN FEET; BILATERAL (Nervous system disorders) | 1
Other, Specify: FOREHEAD NUMBNESS. POST INJECTION #1. (Nervous system disorders) | 1
Other, Specify: INTRACRANIAL ANEURYSM, NONRUPTURED (Nervous system disorders) | 1
Other, Specify: L HEMIPARESIS (Nervous system disorders) | 1
Other, Specify: L SIDED NEGLECT (Nervous system disorders) | 1
Other, Specify: NIGHTMARES (Nervous system disorders) | 1
Other, Specify: PSEUDOMENINGOCELE (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 7
Peripheral sensory neuropathy (Nervous system disorders) | 1
Pyramidal tract syndrome (Nervous system disorders) | 2
Seizure (Nervous system disorders) | 8
Tremor (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 3
Confusion (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 4
Hallucinations (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 4
Restlessness (Psychiatric disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Other, Specify: "PASSING AIR WHEN URINATING" (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Urinary urgency (Renal and urinary disorders) | 1
Other, Specify: LUMP IN LEFT BREAST (Reproductive system and breast disorders) | 1
Testicular pain (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Other, Specify: CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Scalp pain (Skin and subcutaneous tissue disorders) | 1
Other, Specify: FLUID FILLED POCKET ON R FOREHEAD FROM SURGERY (Skin and subcutaneous tissue disorders) | 1
Other, Specify: FLUID POCKET (Skin and subcutaneous tissue disorders) | 1
Other, Specify: RASH (Skin and subcutaneous tissue disorders) | 1
Other, Specify: RIGHT LOWER EXTREMITY. SKIN DISCOLORATION. (Skin and subcutaneous tissue disorders) | 1
Other, Specify: SKIN BUMP (Skin and subcutaneous tissue disorders) | 1
Other, Specify: SKIN SLOUGHING (Skin and subcutaneous tissue disorders) | 1
Skin induration (Skin and subcutaneous tissue disorders) | 17
Hypertension (Vascular disorders) | 24
Thromboembolic event (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-11): https://cdn.clinicaltrials.gov/large-docs/47/NCT02193347/Prot_SAP_000.pdf